CLINICAL TRIAL: NCT01333501
Title: A 18-month, Open-label, Rater-blinded, Randomized, Multi-center, Active-controlled, Parallel-group Pilot Study to Assess Efficacy and Safety of Fingolimod in Comparison to Interferon Beta 1b in Treating the Cognitive Symptoms Associated to Relapsing-remitting Multiple Sclerosis and to Assess Possible Relationship of These Effects to Regional Brain Atrophy
Brief Title: Fingolimod Versus Interferon Beta 1b in Cognitive Symptoms
Acronym: Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DIT01; 2010-023023-19 (EudraCT Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; cognitive symptoms; relapsing-remitting multiple sclerosis (RRMS); fingolimod; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Multiple Sclerosis; Neurobehavioral Manifestations; Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride; Interferon beta-1b

ARMS (2):
- Fingolimod (Experimental): 0.5 mg in capsules for oral administration once daily
  Interventions: Drug: Fingolimod
- Interferon beta 1b (Active Comparator): 250 μg injected s.c. every other day
  Interventions: Drug: Interferon beta 1b

INTERVENTIONS:
Drug: Fingolimod — 0.5 mg in capsules for oral administration once daily
  Arms: Fingolimod
Drug: Interferon beta 1b — 250 μg injected s.c. every other day
  Arms: Interferon beta 1b

SUMMARY:
The purpose of this pilot study is to evaluate, by means of a specific cognitive test battery (Brief Repeatable Battery and Delis-Kaplan Executive Function System scale), the slowing/reduction of cognitive dysfunction progression in RRMS patients after 18 months of treatment with fingolimod in comparison with interferon beta 1b treatment, and to evaluate which test of the battery is the most sensitive in detecting differences between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting forms of MS defined by 2005 revised McDonald criteria.
* Patients with active disease, defined as at least one clinical relapse in the last year, or two clinical relapses in the last two years if there are signs of disease activity at one brain MRI scan performed in the last six months.
* Patients with cognitive impairment at screening, defined as at least one test of the Rao's Brief Repeatable Battery with scores falling outside the 90th percentile of the normative data.

Exclusion Criteria:

* Patients who had already been treated with multiweekly interferon (interferon beta 1b, or beta 1a multiweekly) and had an unsatisfactory response according to the judgment of the investigator.
* Patients with hyperactive forms of the MS disease according to the judgment of the investigator.
* Patients with an EDSS score higher than 5.
* Patients with a prior or current diagnosis of Major Depression according to DSM-IV.
* Patients with a history of chronic disease of the immune system other than MS such as known immunodeficiency syndrome.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Germany (4):
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Würzburg
- Italy (16):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Cefalù, PA
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Gallarate, VA
  - Novartis Investigative Site, Napoli

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total patients randomized in the study (157). Patients who took at least one dose of study drug are 151. The study there were 6 patients who were enrolled but who never took any dose of study drug.
Period: Overall Study
Arm/Group | Fingolimod | Interferon Beta 1b
Started | 106 | 51
Full Analysis Set (FAS) | 80 | 28
Safety Population | 104 | 47
Completed | 97 | 30
Not Completed | 9 | 21
Not completed — Adverse Event | 3 | 1
Not completed — Abnormal laboratory value | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 7
Not completed — Withdrawn consent | 3 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Interferon Beta 1b | Total
Number analyzed (Participants) | 104 | 47 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.53 (9.28) | 37.53 (9.27) | 38.91 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 30 | 98
  Male | 36 | 17 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Screening in Selective Reminding Test - Long-Term Storage (SRT-LTS) Raw Score
Description: Brief Repeatable Battery (BRB)- widely used as a clinical and research tool, with 68% sensitivity and 85% specificity. It consists of the serial administration of 5 tests. One of the tests is SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total of the words in LTS of all six trials is then summed. The total score ranged from 0 to 72. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: Full analysis set (FAS) - all randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of both primary efficacy variables (i.e. non-missing information about the BRB and DKEFS - Sorting test) without any major protocol violations.
Measure: Least Squares Mean (Standard Error); unit: raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
raw score | 6.32 (1.33) | 4.46 (2.28)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.4940, ANCOVA; Mean Difference (Net) = 1.86, 95% CI 2-sided [-3.51 to 7.23], Standard Error of Mean 2.70

2. Primary Outcome: Change From Screening in Selective Reminding Test - Consistent Long Term Retrieval (SRT-CLTR) Raw Score
Description: Brief Repeatable Battery (BRB)- widely used as a clinical and research tool, with 68% sensitivity and 85% specificity. It consists of the serial administration of 5 tests. One of the tests is SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total of the words in LTS of all six trials is then summed. If a word in LTS is consistently recalled on all subsequent trials, it is then scored as Consistent Long Term Retrieval (CLTR). The total of the words in CLTR of all six trials is summed. The total score ranged from 0 to 72. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 5.93 (1.49) | 3.96 (2.56)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.5183, ANCOVA; Mean Difference (Net) = 1.97, 95% CI 2-sided [-4.06 to 7.99], Standard Error of Mean 3.03

3. Primary Outcome: Change From Screening in Spatial Recall Test (SPART) Raw Score
Description: Spatial Recall Test (SPART) for visuospatial learning and delayed recall.Spatial Recall Test (10/36): The spatial recall test assesses visuospatial learning and delayed recall (10/36-D). A checkerboard with ten checkers arranged in a pattern is shown to the subject for ten seconds. The subject is then asked to reproduce the same pattern with ten checkers on an empty checkerboard. The test includes three consecutive trials. The score is the total number of correct responses for the tree trials. The total score ranged from 0 to 30. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 1.46 (0.52) | 3.06 (0.89)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.1334, ANCOVA; Mean Difference (Net) = -1.60, 95% CI 2-sided [-3.69 to 0.50], Standard Error of Mean 1.05

4. Primary Outcome: Change From Screening in Symbol Digit Modalities Test (SDMT) Raw Score
Description: Symbol Digit Modality Test (SDMT) for sustained attention and information processing speed. It presents a series of nine symbols, each of which is paired with a single digit labeled 1-9 in a key at the top of the sheet. The reminder of the page has a pseudo-randomized sequence of symbols, and the patient must respond with the digit associated with each of these as quickly as possible. The score is the number of correct answers in 90 seconds. The total score ranged from 0 to 110. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 2.19 (1.12) | 3.93 (1.93)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.4501, ANCOVA; Mean Difference (Net) = -1.73, 95% CI 2-sided [-6.27 to 2.81], Standard Error of Mean 2.29

5. Primary Outcome: Change From Screening in Paced Auditory Serial Addition Test - 3 Seconds (PASAT 3) Raw Score
Description: Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The patient hears a series of numbers from recordings that are presented at the rate of one every 3 seconds in the first part of the test (PASAT-3). The patient is asked to add each consecutive digit to the one immediately preceding it. Sixty-one digits are presented for each part, and each part has a maximum of 60 correct answers. The total score ranged from 0 to 60. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 7.14 (1.24) | 6.68 (2.13)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.8561, ANCOVA; Mean Difference (Net) = 0.46, 95% CI 2-sided [-4.57 to 5.49], Standard Error of Mean 2.53

6. Primary Outcome: Change From Screening in Paced Auditory Serial Addition Test - 2 (PASAT 2) Raw Score
Description: Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The patient hears a series of numbers from recordings that are presented at the rate of one every 2 seconds in the second part of the test (PASAT-2). The patient was asked to add each consecutive digit to the one immediately preceding it. Sixty-one digits are presented for each part, and each part has a maximum of 60 correct answers. The total score ranged from 0 to 60. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 4.79 (1.25) | 4.42 (2.14)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.8858, ANCOVA; Mean Difference (Net) = 0.37, 95% CI 2-sided [-4.67 to 5.40], Standard Error of Mean 2.53

7. Primary Outcome: Change From Screening in Selective Reminding Test - Delayed Recall (SRT-D) Raw Score
Description: The tests SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall). The Delayed SRT test is the total number of words recalled after a delayed period. The total score ranged from 0 to 12. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 0.57 (0.23) | 0.39 (0.40)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.7119, ANCOVA; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.76 to 1.11], Standard Error of Mean 0.47

8. Primary Outcome: Change From Screening in Spatial Recall Test - Delayed Recall (SPART-D)
Description: Spatial Recall Test (SPART) for visuospatial learning and delayed recall.Spatial Recall Test (10/36): The spatial recall test assesses visuospatial learning and delayed recall (10/36-D). A checkerboard with ten checkers arranged in a pattern was shown to the subject for ten seconds. The subject was then asked to reproduce the same pattern with ten checkers on an empty checkerboard. The test includes three consecutive trials. The score was the total number of correct responses for the tree trials. The total score ranged from 0 to 10. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 0.41 (0.21) | 0.44 (0.36)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.9496, ANCOVA; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.86 to 0.81], Standard Error of Mean 0.42

9. Primary Outcome: Change From Screening in Word List Generation (WLG)
Description: Word List Generation (COWAT/WLG): The COWAT assesses verbal fluency on semantic stimulus by asking the patient to produce as many words as possible belonging to a semantic category. The test assessed the verbal fluency, recorded all the possible correct word that a patients should give in 90 sec. No maximum range is available. Higher values represent a better outcome. The score was the number of correct words. The more words the patient pronounces, the better it is. We can imagine that the minimum value might be zero words, , but it is not a score scale.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 0.39 (0.58) | 0.24 (0.99)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.8944, ANCOVA; Mean Difference (Net) = 0.16, 95% CI 2-sided [-2.18 to 2.50], Standard Error of Mean 1.18

10. Primary Outcome: Change From Screening in Delis-Kaplan Executive Function System (DKEFS) Condition 1: Free Sorting, Confirmed Correct Sort- Card Set 1+2
Description: The Delis-Kaplan Executive Function System - Sorting Test is one of the nine tests presented in the DKEFS manual and explores the patient's executive abilities. It has a standard form (version A, administered at screening and Month-18 visit) and an alternate form (version B, administered at Month-9 visit). The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. The DKFES test consisted of two testing procedures: free sorting and sort recognition. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) was obtained, as well as the sum of description scores of both sets. The total score ranged from 0 to 16. Higher values represent a better outcome
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 0.57 (0.31) | 0.82 (0.48)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.6757, ANCOVA; Mean Difference (Net) = -0.25, 95% CI 2-sided [-1.42 to 0.92], Standard Error of Mean 0.59

11. Primary Outcome: Change From Screening in DKEFS Condition 1: Free Sorting, Free Sorting, Description Score, Card Set 1+2
Description: The Delis-Kaplan Executive Function System - Sorting Test is one of the nine tests presented in the DKEFS manual and explores the patient's executive abilities. It has a standard form (version A, administered at screening and Month-18 visit) and an alternate form (version B, administered at Month-9 visit). The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) was obtained, as well as the sum of description scores of both sets. The total score ranged from 0 to 64. Higher values represent a better outcome
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 1.52 (1.23) | 3.69 (1.92)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.3585, ANCOVA; Mean Difference (Net) = -2.16, 95% CI 2-sided [-6.82 to 2.50], Standard Error of Mean 2.34

12. Primary Outcome: Change From Screening in DKEFS Condition 2: Sort Recognition, Sort Recognition Description Score- Card Set 1+2
Description: The Delis-Kaplan Executive Function System - Sorting Test is one of the nine tests presented in the DKEFS manual and explores the patient's executive abilities. It has a standard form (version A, administered at screening and Month-18 visit) and an alternate form (version B, administered at Month-9 visit). The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. Free sorting and sort recognition. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. The total score ranged from 0 to 64. Higher values represent a better outcome.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | 2.15 (1.90) | 7.38 (2.97)
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta 1b; Test type: Superiority or Other; p = 0.1610, ANCOVA; Mean Difference (Net) = -5.24, 95% CI 2-sided [-12.62 to 2.14], Standard Error of Mean 3.69

13. Secondary Outcome: Change From Screening in the Volume of Total T2 Lesions
Description: Change in volume of total T2-weighted lesions by visit were summarized. Negative values indicate improvement (reduction in lesion volume) and positive values worsening (increase in lesion volume
Time Frame: Screening (-1 month), 18 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 68 | 27
mm^3 | 176.25 (1355.31) | 711.81 (1584.42)

14. Secondary Outcome: Change From Screening in Montgomery-Asberg Depression Rating Scale (MADRS)
Description: MADRS measures the overall severity of depressive symptoms. The MADRS had a 10-item checklist. Items are rated on a scale of 0-6, for a total numeric range of scores from 0 (depressive symptoms absent) to 60 (numerically highest level of depressive symptoms).
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Raw score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Raw score | -0.77 (0.79) | 0.13 (1.31)

15. Secondary Outcome: Changes in Quality of Life, by Means of the Multiple Sclerosis Quality of Life (MSQoL-54)
Description: A 54 question measure covers 12 domains; assesses mental and physical health. The physical health composite score is a weighted average of the physical health scales, such as physical function, health perceptions, and energy. The mental health composite score is a weighted average of the mental health scales, such as overall quality of life, cognitive function, and health distress. Each domain has a range from 0 to 100 where higher means better.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Score
  Mental health composite score | 4.76 (2.01) | -2.31 (3.36)
  Physical health composite score | -1.80 (1.41) | -4.75 (2.46)

16. Secondary Outcome: Changes From Baseline in Fatigue Impact Scale (mFIS, Total Score and Scores of the 3 Individual Domains).
Description: Modified Fatigue Impact Scale (mFIS) questionnaire is described at each time point to evaluate fatigue by means of usual descriptive statistics. Three domains were also defined: Physical Subscale (sum of items 4, 6, 7, 10, 13, 14, 17, 20, 21 and therefore ranging from 0 to 36), Cognitive Subscale (sum of items 1, 2, 3, 5, 11, 12, 15, 16, 18, 19 and therefore ranging from 0 to 40) and Psychosocial Subscale (sum of items 8, 9 and therefore ranging from 0 to 8). Finally, mFIS - overall score ranged from 0 to 80. The mFIS total score was computed as the sum of scores for each item. Lower values represent a better outcome.
Time Frame: Baseline, 18 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Score | 2.36 (1.68) | 6.67 (2.72)

17. Secondary Outcome: Change From Screening in the Number of New T2 Lesions
Description: New T2 lesions at a specific visit were assessed relative to the previous visit scan. The total number of lesions (visit 8 to 18 month) is calculated as the sum of the number of lesions.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of new lesions
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Number of new lesions | 1.25 (2.05) | 3.33 (4.44)

18. Secondary Outcome: Change From Screening in the Volume of Total T1 Hypointense Lesions
Description: Volume of hypointense post-gadolinium T1 lesion component was measured by MRI scan. Means were estimated using a Mixed-effect model with repeated measures (MMRM) by-visit interaction.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
mm^3 | 391.96 (986.85) | 213.93 (312.24)

19. Secondary Outcome: Change From Screening in the Number of T1 Gd+ Enhancing Lesions
Description: Total number of post-baseline Gd-enhanced lesions is calculated as a sum of all Gd-enhanced lesions seen on post-baseline scans per visit. Real (not per slice) lesions are counted in this analysis
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of new lesions
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Number of new lesions | -0.64 (1.27) | 0.59 (3.98)

20. Secondary Outcome: Change From Screening in the Percentage of Brain Volume Change
Description: Calculations of brain volume change were performed using the structural image evaluation of normalized atrophy (SIENA), software included in the Functional Magnetic Resonance Imaging of the Brain (FMRIB) software library. SIENA is a fully automated method for estimating temporal brain volume change.
Time Frame: Screening (-1month), 18 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of brain volume
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
percentage of brain volume | -0.60 (0.83) | -0.96 (0.71)

21. Secondary Outcome: Changes in the Environmental Status Scale Score (ESS)
Description: The Environmental Status Scale (ESS) is used to quickly evaluate a patient for handicap. It was derived from a measure of socio-economic status. It consists of seven parameters: (1) actual work status, (2) financial and economic status, (3) personal residence or home, (4) personal assistance required, (5) transportation, (6) community services, (7) social activity. Each parameter has a single score from minimum 0 to maximum 5. ESS score is the sum of the points for all 7 parameters: minimum score: 0; maximum score: 35. The higher the score the greater the handicap
Time Frame: Baseline, 18 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Fingolimod | Interferon Beta 1b
Number analyzed (Participants) | 80 | 28
Score | 1.08 (3.45) | 0.91 (1.98)

ADVERSE EVENTS:
Groups:
- Fingolimod 0.5 mg: 0.5 mg in capsules for oral administration once daily
Arm/Group | Fingolimod 0.5 mg | Interferon Beta 1b
Serious Adverse Events (participants affected / at risk) | 9/104 | 1/47
Other Adverse Events (participants affected / at risk) | 44/104 | 22/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=104) | Interferon Beta 1b (N=47)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose abnormal (Investigations) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Uterine polypectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=104) | Interferon Beta 1b (N=47)
Influenza like illness (General disorders) | 1 | 5
Pyrexia (General disorders) | 6 | 4
Nasopharyngitis (Infections and infestations) | 4 | 3
Alanine aminotransferase increased (Investigations) | 9 | 1
Blood triglycerides increased (Investigations) | 0 | 3
Transaminases increased (Investigations) | 4 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 11 | 4
Multiple sclerosis relapse (Nervous system disorders) | 2 | 4
Depression (Psychiatric disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.